CLINICAL TRIAL: NCT05433649
Title: Effects of Therapeutic Exercise With Elastic Bands on Strength and Pain in Women With Non-specific Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Pablo Hernandez-Lucas, Associate professor in health sciences, University of Vigo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0004
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Neck Pain; Exercise Therapy; Women
MeSH Terms: conditions — Neck Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants performing 16 sessions of therapeutic exercise for 8 weeks with a frequency of two sessions per week. All sessions had a practical focus (strength and stretching exercises) with the help of elastic bands.
  Interventions: Behavioral: Therapeutic exercise
- Control group (No Intervention): They do not change their lifestyle and do not receive the therapeutic exercise sessions.

INTERVENTIONS:
Behavioral: Therapeutic exercise — The therapeutic exercise intervention with the help of elastic bands was carried out for 8 weeks with a frequency of two sessions per week, for a total of 16 sessions of 45 minutes duration.
  Arms: Experimental group

SUMMARY:
The study consists of an intervention of 16 therapeutic exercise sessions during 8 weeks with a frequency of two sessions per week. All sessions had a practical focus (strength and stretching exercises) with the help of elastic bands. In addition, they had an initial session and another at the end of the intervention in which measurements of the different variables (cervical pain, cervical flexor strength, cervical extensor strength and strength of the scapular stabilising musculature) were taken on two occasions, at the beginning of the study and at the end of the intervention, an average of 2 months.

Nonspecific neck pain has a higher incidence in women than in men. Female sex is a risk factor for this pathology. Clinical practice guidelines highlight the importance of preventing neck pain through exercise. There are previous studies on the effects of strength programmes on patients with non-specific neck pain, but none have used elastic bands as an implement, despite the fact that it is one of the most commonly used implements in physiotherapy clinics. Therefore, the aim of this study is to investigate the effects of an elastic band therapeutic exercise intervention in women with non-specific neck pain. It was previously hypothesised that this intervention would have positive effects on pain and strength in the cervical and scapular region.

ELIGIBILITY:
Inclusion Criteria:

* Women.
* 18-65 years of age.
* With non-specific neck pain for at least three months, with pain intensity (30-70 on a VAS).

Exclusion Criteria:

* Any previous neck or shoulder surgery, fibromyalgia, cervical radiculopathy/myelopathy, history of the whiplash injury, cognitive disorder.
* Missing more than sessions.
* Not being able to attend the measurement sessions.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Through study completion, an average of 2 months
  The visual analogue scale is a widely used tool for measuring pain. The patient is asked to indicate their perceived pain intensity (most commonly) along a 100 mm horizontal line, and this rating is then measured from the left edge. With 0 mm being no pain perception and 100 mm being the maximum perceived pain. So the higher the value the worse the patient's pain sensation.
Neck flexor muscle endurance. | Through study completion, an average of 2 months
  This was measured using the deep neck flexor endurance test. When in supine position, participants were asked to flex the upper cervical spine, move their heads away from the couch approximately 2.5 cm and hold this position for as long as possible. The test ended when students dropped their heads or lost craniocervical flexion.
Neck extensor muscle endurance. | Through study completion, an average of 2 months
  Students were in prone position, head neutral, arms by their sides and a 10-cm stabilising strip of Velcro was placed at the sixth dorsal vertebra level. An inclinometer and 5-cm strap were placed around the participants head with a 2-kg weight hanging from it. Participants were asked to support this weight for as long as possible while maintaining a neutral head position.
Scapular stabiliser endurance. | Through study completion, an average of 2 months
  Participants stood with their shoulders and elbows flexed at 90°. Students' elbows were kept approximately shoulder-distance apart with a ruler and they were asked to pull both extremities of the dynamometer by externally rotating their shoulders until the dynamometer reached 1 kg. They were asked to hold this position for as long as possible.

CONTACTS AND LOCATIONS:
Locations (1):
- Pablo Hernández Lucas, Pontevedra, Spain

REFERENCES:
- [Derived] Hernandez-Lucas P, Leiros-Rodriguez R, Lopez-Barreiro J, Garcia-Soidan JL. Effects of exercise therapy using elastic bands on strength and pain in women with non-specific neck pain: A randomised controlled trial. Heliyon. 2023 Nov 14;9(11):e22237. doi: 10.1016/j.heliyon.2023.e22237. eCollection 2023 Nov. PMID 38058646